CLINICAL TRIAL: NCT02445027
Title: Pilot Study for Imaging of the Esophagus Using a Tethered Capsule OCT Endomicroscopy in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014-P001519
Record Dates: First submitted 2015-02-26; First posted 2015-05-15 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Primary Care; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MGH OCT Imaging Capsule (Experimental): Subject will swallow the OCT capsule and images will be acquired using the OCT Imaging system.
  Interventions: Device: MGH OCT Imaging Capsule

INTERVENTIONS:
Device: MGH OCT Imaging Capsule — Imaging of the esophagus using the OCT Capsule and system.

SUMMARY:
The goal of this study is to test the feasibility and acceptability of tethered capsule Optical Coherence Tomography (OCT) endomicroscopy as a device for population-based screening in the primary care practice environment.

DETAILED DESCRIPTION:
60 healthy volunteers scheduled for a routine primary care visit will be recruited and asked to swallow the OCT capsule while being awake and unsedated. The capsule is attached to a tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus using natural propulsive force called peristalsis.

As the capsule progresses through the esophagus, multiple images of the esophagus are acquired and later analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be scheduled for non-urgent appointment at primary care practice including annual wellness visits and routine follow-up appointments.
* Subjects must be over the age of 18
* Subjects must be able to give informed consent
* Subjects must have no solid food for 4 hours prior to the procedure, and only clear liquids for 2 hours prior to the procedure.

Exclusion Criteria:

* Subjects with current symptoms of dysphagia
* Subjects with any history of intestinal strictures, prior GI surgery, or history of intestinal Crohn's disease.
* Subjects with current symptoms of fever, nausea or sore throat at the time of the appointment.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total number of 60 Participants were enrolled in the study
Groups:
- Feasibility of Tethered Capsule Endomicroscopy: Number of participants able to swallow the capsule and capture OCT images successfully in the PCP setting.
Period: Overall Study
Arm/Group | Feasibility of Tethered Capsule Endomicroscopy
Started | 60
Completed | 45
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Feasibility: Number of participants able to swallow the capsule and capture OCT images successfully.
Arm/Group | Feasibility
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 49
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Esophageal Imaging in Subjects Who Successfully Swallow the OCT Capsule in the Primary Care Setting.
Description: Number of Participants able to swallow the capsule successfully. An investigator will assess the quality of the recorded images and movies obtained with each exam after imaging has been completed. This is a feasibility study and was not used for any diagnosis.
Time Frame: Approximate 20min visit (5min image acquisition)
Measure: Count of Participants; unit: Participants
Groups:
- Feasibility: Feasibility is measured by the total number of Participants able to swallow the capsule successfully.
Arm/Group | Feasibility
Number analyzed (Participants) | 60
Participants | 45

ADVERSE EVENTS:
Time Frame: During the procedure and 10 minutes after
Description: The adverse events were collected systematically for this study. The definition of adverse events is the same as clinicaltrials.gov definition.
Arm/Group | MGH OCT Imaging Capsule
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT02445027/Prot_SAP_000.pdf